CLINICAL TRIAL: NCT06876688
Title: Relmacabtagene Autoleucel Injection Followed by Tislelizumab for the Treatment of Relapsed/Refractory Large B-Cell Lymphoma Involved in the Central Nervous System
Brief Title: Relma-cel Followed by Tislelizumab for the Treatment of Relapsed/Refractory CNS Large B-Cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNSL-CART
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: CNS Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention group (Experimental): Relma-cel Followed by Tislelizumab
  Interventions: Drug: Relma-cel Followed by Tislelizumab

INTERVENTIONS:
Drug: Relma-cel Followed by Tislelizumab — Enrolled patients with relapsed/refractory (R/R) CNSL will receive Relma-cel infusion, followed by treatment with Tislelizumab (200mg, IV, q4w, for 12 months) starting at 35 days post-infusion. BTK inhibitors will be used in combination as needed.

SUMMARY:
This study aims to evaluate the efficacy and safety of Relma-cel in the treatment of central nervous system lymphoma (CNSL), as well as its pharmacokinetic characteristics. Enrolled patients with relapsed/refractory (R/R) CNSL will receive Relma-cel infusion, followed by Tislelizumab treatment (200mg, IV, q4w, for 12 months) starting on day 35 after infusion. Bruton's tyrosine kinase (BTK) inhibitors will be used in combination as needed. The follow-up period will last for 4 years, monitoring drug safety, disease status, survival, and the pharmacokinetic characteristics of Relma-cel.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 18 years old, male or female;
2. Relapsed or refractory CNS-involved large b-cell lymphoma after at least first-line therapy, with an efficacy assessment of CR or PR after salvage therapy, and current stable efficacy status;
3. Eastern Cooperative Oncology Group (ECOG) score of 0-2;
4. Have a life expectancy of ≥ 12 weeks
5. Use contraception
6. Have adequate bone marrow and organ function:

   1. Neutrophil count (anc) ≥1.0 x 109/L;
   2. Hemoglobin ≥ 8.0 g/dl;
   3. Platelet count ≥ 50 x 109/L;
   4. Total bilirubin ≤ 1.5 × upper limit of normal (ULN)
   5. Alanine aminotransferase/aspartate aminotransferase (ALT/AST) ≤ 2.5 x ULN or ≤ 5 x ULN (in the presence of hepatic invasion);
   6. Creatinine clearance ≥40mL/min
   7. Lipase ≤ 1.5 x ULN

Exclusion Criteria:

1. Severe active central nervous system symptoms
2. Prior chimeric antigen receptor cellular immunotherapy targeting cd19
3. Known human immunodeficiency virus (hiv) infection or positive immunoassay;
4. Live vaccination within 30 days prior to study drug administration;
5. Active autoimmune disease requiring systemic therapy in the last 12 months
6. Allergy to the study drug or history of severe allergic reactions
7. Potential risk of malignant cardiac arrhythmia
8. History of stroke or intracranial hemorrhage within 3 months prior to the date of administration of study medication
9. Other malignant tumors presently or within 3 years prior to enrollment
10. Conditions that, in the judgment of the investigator, would interfere with full participation in the study; pose a significant risk to the subject; or interfere with the interpretation of the study data
11. Pregnant or lactating patients;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Complete response rate(CRR) at 3-month | 3 months post CAR-T infusion
  Complete response rate at 3-month is defined as the incidence of subjects achieving complete response (CR) at 3-month after CAR-T infusion according to the Lugano Classification, as determined by study investigators.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | 2 years post CAR-T infusion
  PFS is defined as the time from the CAR-T infusion date to the date of disease progression or death from any cause.
Overall Survival (OS) | 2 years post CAR-T infusion
  OS is defined as the time from CAR-T infusion to the date of death from any cause.
Objective remission rate (ORR) at 3-month | 3 months post CAR-T infusion
  Objective remission rate (ORR) at 3-month is defined as the incidence of either a CR or a partial response (PR) at 3-month after CAR-T infusion per the Lugano Classification as determined by study investigators

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Beljing Tiantan Hospital, Capttal Medical, University, Beijing
  - Xuanwu Hospital Capital Medical University, Beijing
  - Sun Yat-Sen University Cancer Center, Guangzhou
  - Henan Cancer Hospital, Henan
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology,, Wuhan